CLINICAL TRIAL: NCT05636423
Title: Sexual Disability Related to Low Back Pain. Online Survey Among Italian Physiotherapists.
Brief Title: Sexual Disability in Low Back Pain and Physiotherapy
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Paolo Pillastrini, Full Professor, University of Bologna
Other Study IDs: Sex and LBP
Record Dates: First submitted 2022-11-16; First posted 2022-12-05 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Low Back Pain; Sex Disorder
Keywords: sexual disability; physical therapy; low back pain
MeSH Terms: conditions — Low Back Pain; Sexual Dysfunction, Physiological | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Italian physiotherapists: The survey will take place through the administration of a questionnaire accessible via the website of the Italian Physiotherapy Association (AIFI), the Scientific Association of reference for the physiotherapists, registered since 2020 in the list of Scientific Societies recognized by the Italian Health Ministry.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Online survey via a questionnaire composed of 28 questions.

SUMMARY:
A treatment centered on the person uses an approach capable of considering all the components of disability, from a physical, psychological and social point of views. Some studies have shown that sexual function is disturbed in subjects with low back pain (LBP) and sexual disability can contribute to a deterioration in quality of life. It has also been shown that, in sexually active patients complaining of LBP, sexuality is a significant mediator of the relationship between pain intensity and depressive symptoms.

The Oswestry Disability Index (ODI) includes a specific item to investigate sexual function (item #8). A previous study of ours confirmed the relationship between sexual disability detected by the ODI and the presence of depression, avoidance of activities and rumination (Ferrari et al. 2019 - Digital Object Identifier: 10.1589/jpts.31.360).

The discussion on sexual disability among patients and healthcare professionals is very limited, although patients require more involvement from clinicians, especially physiotherapists, as evidenced by our previous qualitative study (Ferrari et al. 2020 - Digital Object Identifier: 10.1080/09638288.2020 .1817161).

Although studies on this topic have highlighted the importance of this disability in the life of subjects complaining of LBP, little has been investigated on clinical behaviors of the physiotherapists in this area.

DETAILED DESCRIPTION:
The goal of this observational study is to learn about the clinical behaviors of Italian physiotherapists in the management of LBP-related sexual disability. The main questions it aims to answer are:

* the knowledge of this topic;
* the ways in which sexual disability is detected in patients complaining of LBP (Oswestry Disability Index, specific open or closed questions, patient' reporting, etc.);
* the difficulties and obstacles in the management of sexual disability;
* the suggestions provided to the patient;
* the therapeutic strategies (procedures for pain modulation, exercises addressed to lumbar mobility, strength, endurance, etc.);
* the possible involvement of the patient' partner;
* the outcome measures.

The hypothesis of this survey is to highlight the degree of attention and competence of Italian physiotherapists with respect to this topic, the critical issues and therapeutic strategies for the management of LBP-related sexual disability.

Participants will answer to a online questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Being a physiotherapist registered with AIFI
* Carrying out physiotherapy treatments on subjects with low back pain
* Agreement to voluntarily sign informed consent to participate in the study
* Agreement to voluntarily sign consent to data processing

Exclusion Criteria:

* Inability to understand written Italian
* Being a retired physiotherapist

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physiotherapists registered with AIFI who deliver physiotherapy treatments on subjects with low back pain
Sampling Method: Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-06-24 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Clinical behaviors of Italian physiotherapists regarding sexual disability in patients with low back pain | From date of first completion of the survey until the date of last completion of the survey.
  Level of attention and competence of Italian physiotherapists with respect to sexual disability related to low back pain, critical issues, opportunities and therapeutic strategies adopted in the management of sexual disability related to LBP.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pillastrini, PT, MSc, Principal Investigator — University of Bologna
Locations (1):
- Policlinico S. Orsola-Malpighi, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrari S, Vanti C, Giagio S, Anesi M, Youssef S, Bortolami A, Cedraschi C, Pillastrini P. Low back pain and sexual disability from the patient's perspective: a qualitative study. Disabil Rehabil. 2022 May;44(10):2011-2019. doi: 10.1080/09638288.2020.1817161. Epub 2020 Sep 15. PMID 32931339
- [Background] Ferrari S, Vanti C, Frigau L, Guccione AA, Mola F, Ruggeri M, Pillastrini P, Monticone M. Sexual disability in patients with chronic non-specific low back pain-a multicenter retrospective analysis. J Phys Ther Sci. 2019 Apr;31(4):360-365. doi: 10.1589/jpts.31.360. Epub 2019 Apr 1. PMID 31037010